CLINICAL TRIAL: NCT01896479
Title: A Randomized, Double-blind Study To Evaluate the Efficacy and Safety of Cabozantinib (XL184) at 60 mg/Day Compared to a 140 mg/Day in Progressive, Metastatic Medullary Thyroid Cancer Patients
Brief Title: A Study of Two Different Doses of Cabozantinib (XL184) in Progressive, Metastatic Medullary Thyroid Cancer
Acronym: EXAMINER
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL184-401; 2024-516480-90-00 (EU CTIS Number)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Medullary Thyroid Cancer
Keywords: thyroid cancer; medullary thyroid cancer
MeSH Terms: conditions — Carcinoma, Medullary; Thyroid Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabozantinib (XL184) 60 mg (Experimental): Cabozantinib (XL184) 140 mg as capsules and placebo tablets administered orally once a day.
  Interventions: Drug: Cabozantinib (XL184) 60 mg; Drug: Placebo capsule
- Cabozantinib (XL184) 140 mg (Experimental): Cabozantinib (XL184) 140 mg as tablets and placebo capsules administered orally once a day.
  Interventions: Drug: Cabozantinib (XL184) 140 mg; Drug: Placebo tablet

INTERVENTIONS:
Drug: Cabozantinib (XL184) 140 mg
  Arms: Cabozantinib (XL184) 140 mg
Drug: Cabozantinib (XL184) 60 mg
  Arms: Cabozantinib (XL184) 60 mg
Drug: Placebo tablet
  Arms: Cabozantinib (XL184) 140 mg
Drug: Placebo capsule
  Arms: Cabozantinib (XL184) 60 mg

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of oral cabozantinib at a 60 mg dose compared with a 140 mg dose in subjects with progressive, metastatic MTC. It will test if the lower dose results in similar progression free survival (PFS) and overall response rate (ORR) with fewer adverse events compared to the PFS, ORR and adverse events found in previous clinical trials of 140 mg.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a histologically confirmed diagnosis of MTC.
2. All subjects will need to be tested for RET mutational status. If subjects do not have documentation confirming they have a RET mutation, a sample of their tumor (taken either during screening or from a procedure within 6 months prior to randomization) will need to be tested.
3. The subject has measurable disease per RECIST 1.1 that is metastatic as determined by the investigator based upon computerized tomography (CT), magnetic resonance imaging (MRI), PET scan, bone scan, or X-ray taken within 28 days before randomization.
4. The subject has documented worsening of disease (progressive disease) at screening as compared with a previous CT, PETor MRI scan, bone scan, or X-ray as determined by the investigator per RECIST 1.1 on qualifying screening images taken within 28 days prior to randomization as compared to previous images taken within 14 months before the qualifying screening images.
5. The subject has recovered to baseline or CTCAE v4.0 (Common Terminology Criteria for Adverse Events, version 4.0) ≤ Grade 1 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
6. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 at screening.
7. The subject has adequate organ and marrow function
8. The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document.
9. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (eg, barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment.

Exclusion Criteria:

1. The subject has previously received cabozantinib.
2. Receipt of any type of small molecule kinase inhibitor or hormonal therapy within 28 days or 5 half-lives of the compound or active metabolites, whichever is shorter, before randomization.
3. Receipt of any systemic anti-tumor therapy within 28 days of randomization (42 days for nitrosoureas or/ mitomycin C).
4. Receipt of any other type of investigational agent within 28 days of randomization.
5. Receipt of radiation therapy within 28 days (14 days for radiation for bone metastases) of randomization or radionuclide treatment within 42 days of randomization. Subject is ineligible if there are any clinically relevant ongoing complications from prior radiation therapy.
6. The subject has untreated and/or active (progressing or requiring anticonvulsants or corticosteroids for symptomatic control) central nervous system (CNS) metastasis. Must have completed radiation therapy ≥ 28 days prior to randomization and be stable without corticosteroids or anti-convulsant treatment for ≥ 10 days.
7. Treatment at therapeutic doses with oral anticoagulants or platelet inhibitors (examples are warfarin and clopidogrel).
8. The subject has uncontrolled, significant intercurrent illness including, but not limited to, cardiovascular disorders, gastrointestinal disorders, active infections, non-healing wounds, recent surgery.
9. Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before randomization.
10. The subject is unable to swallow multiple tablets or capsules.
11. The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.
12. The subject is pregnant or breastfeeding.
13. The subject has had a diagnosis of another malignancy within 2 years before randomization, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2035-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (45):
- Australia (4):
  - St Leonards, New South Wales
  - Herston, Queensland
  - Kurralta Park, South Australia
  - Parkville, Victoria
- Canada (2):
  - Québec, Quebec
  - Toronto
- Croatia (2):
  - Osijek
  - Zagreb
- France (7):
  - Bordeaux, Gironde
  - Angers, Maine-et-Loire
  - Lyon, Rhône
  - Villejuif, Val-de-Marne
  - Dijon
  - Paris
  - Strasbourg
- Hungary (2):
  - Budapest
  - Debrecen
- Israel (3):
  - Jerusalem
  - Petah Tikva
  - Safed
- Italy (7):
  - Catania, CT
  - Roma, RM
  - Siena, SI
  - Pisa, Tuscany
  - Milan
  - Padua
  - Torino
- Netherlands (3):
  - Amsterdam, North Holland
  - Leiden, South Holland
  - Groningen
- Poland (2):
  - Poznan, Greater Poland Voivodeship
  - Gliwice, Silesian Voivodeship
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Timișoara
- Russia (4):
  - Novosibirsk
  - Obninsk
  - Saint Petersburg
  - Yaroslavl
- South Korea (2):
  - Goyang, Gyeonggido
  - Seoul
- Spain (2):
  - Barcelona
  - Madrid
- Sweden (2):
  - Lund, Skane Ian
  - Uppsala, Uppsala Ian

REFERENCES:
- [Derived] Capdevila J, Klochikhin A, Leboulleux S, Isaev P, Badiu C, Robinson B, Hughes BGM, Keam B, Parnis F, Elisei R, Gajate P, Gan HK, Kapiteijn E, Locati L, Mangeshkar M, Faoro L, Krajewska J, Jarzab B. A Randomized, Double-Blind Noninferiority Study to Evaluate the Efficacy of the Cabozantinib Tablet at 60 mg Per Day Compared with the Cabozantinib Capsule at 140 mg Per Day in Patients with Progressive, Metastatic Medullary Thyroid Cancer. Thyroid. 2022 May;32(5):515-524. doi: 10.1089/thy.2022.0027. PMID 35403447

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cabozantinib-matched placebo capsules and tablets were administered along with the corresponding tablets and capsules to maintain the blinding of the study treatment. Per prespecified analysis, all participants who died during the study met the study requirements of study completion. Therefore, none of the deaths that occurred during the study were recorded as leading to study discontinuation.
Groups:
- Cabozantinib (XL184) 60 mg: Cabozantinib (XL184) 60 milligram (mg) tablets were administered with cabozantinib-matched placebo capsules orally once a day.
- Cabozantinib (XL184) 140 mg: Cabozantinib (XL184) 140 mg capsules were administered with cabozantinib-matched placebo tablets administered orally once a day.
Period: Overall Study
Arm/Group | Cabozantinib (XL184) 60 mg | Cabozantinib (XL184) 140 mg
Started | 123 | 124
Received at Least 1 Dose of Study Drug | 123 | 124
Completed | 123 | 124
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Measured in the Safety Population, which included participants who received any amount of study drug.
Groups:
- Cabozantinib (XL184) 60 mg: Cabozantinib (XL184) 60 mg tablets were administered with cabozantinib-matched placebo capsules orally once a day.
- Total: Total of all reporting groups
Arm/Group | Cabozantinib (XL184) 60 mg | Cabozantinib (XL184) 140 mg | Total
Number analyzed (Participants) | 123 | 124 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 78 | 163
  >=65 years | 38 | 46 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 50 | 83
  Male | 90 | 74 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 103 | 102 | 205
  Unknown or Not Reported | 18 | 16 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 8 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 92 | 102 | 194
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 18 | 13 | 31
Region of Enrollment [Number; unit: participants]
  Romania | 9 | 9 | 18
  Hungary | 4 | 1 | 5
  Russia | 14 | 16 | 30
  Spain | 6 | 12 | 18
  Canada | 2 | 1 | 3
  Netherlands | 4 | 4 | 8
  South Korea | 10 | 7 | 17
  Sweden | 5 | 1 | 6
  Poland | 13 | 17 | 30
  Italy | 9 | 13 | 22
  Israel | 3 | 5 | 8
  Australia | 19 | 20 | 39
  France | 21 | 13 | 34
  Croatia | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Blinded Independent Radiology Committee (BIRC) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS per BIRC per RECIST 1.1 was measured from randomization until the date of first documented disease progression or date of death from any cause, whichever came first, and was assessed for up to 31 months. The prespecified primary analysis was triggered by the required number of at least 150 events occurring in the ITT population, The data cutoff date for this event-driven analysis in the ITT population was when a total of 155 events were reported. Median PFS was calculated using the Kaplan-Meier estimates.
Time Frame: Median time of follow-up (from the date of randomization of the first participant through primary data cut off [15 July 2020]) was 30.2 months
Population: Measured in the Intent-to-Treat (ITT) Population, which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib (XL184) 60 mg | Cabozantinib (XL184) 140 mg
Number analyzed (Participants) | 123 | 124
months | 11 [8.3 to 13.6] | 13.9 [9.0 to 16.6]
Statistical Analysis 1: Comparison: Cabozantinib (XL184) 60 mg vs Cabozantinib (XL184) 140 mg; Test type: Non-Inferiority — The non-inferiority margin used was 1.58; p = 0.1916, Log Rank — Stratification factors comprised RET M918T mutational status (positive, negative, and unknown); Cox Proportional Hazard = 1.24, 95% CI 2-sided [0.90 to 1.70]

2. Secondary Outcome: Objective Response Rate (ORR) Per BIRC Per RECIST 1.1
Description: ORR per BIRC per RECIST 1.1 is the percentage of ITT participants who experienced a best overall response of complete response (CR) or partial response (PR), confirmed ≥ 28 days later, CR defined as disappearance of all non-target lesions. All lymph nodes must have been non-pathological in size (<10 mm short axis). PR defined as unequivocal progression of non-target lesions. Unequivocal progression was to trump target lesion status. It must have been representative of overall disease status change, not a single lesion increase.
Time Frame: as for outcome 1
Population: Measured in the ITT Population, which included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib (XL184) 60 mg | Cabozantinib (XL184) 140 mg
Number analyzed (Participants) | 123 | 124
percentage of participants | 33 [25.09 to 42.40] | 33 [24.88 to 42.08]
Statistical Analysis 1: Comparison: Cabozantinib (XL184) 60 mg vs Cabozantinib (XL184) 140 mg; Test type: Other — Descriptive statistical analysis; p = 0.9437, Cochran-Mantel-Haenszel; Stratification factors comprised RET M918T mutational status (positive, negative, and unknown); Odds Ratio (OR) = 1.0195, 95% CI 2-sided [0.6 to 1.7]

ADVERSE EVENTS:
Time Frame: From first dose to 30 days following last dose (up to a maximum of 61 months)
Description: Measured in the Safety Population, which included participants who received any amount of study drug. Per prespecified analysis, all participants who died during the study met the study requirements of study completion.
Arm/Group | Cabozantinib (XL184) 60 mg | Cabozantinib (XL184) 140 mg
All-Cause Mortality (participants affected / at risk) | 59/123 | 51/124
Serious Adverse Events (participants affected / at risk) | 55/123 | 62/124
Other Adverse Events (participants affected / at risk) | 122/123 | 123/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) 60 mg (N=123) | Cabozantinib (XL184) 140 mg (N=124)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 3
Anal fistula (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Femoral hernia strangulated (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 1 | 2
Death (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 5
Sepsis (Infections and infestations) | 3 | 2
Peritonitis (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Perihepatic abscess (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Amylase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 9
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cerebellar ischaemia (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Aortic dissection rupture (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) 60 mg (N=123) | Cabozantinib (XL184) 140 mg (N=124)
Anaemia (Blood and lymphatic system disorders) | 17 | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 14
Leukopenia (Blood and lymphatic system disorders) | 7 | 15
Lymphopenia (Blood and lymphatic system disorders) | 12 | 10
Neutropenia (Blood and lymphatic system disorders) | 9 | 12
Tachycardia (Cardiac disorders) | 7 | 6
Hypothyroidism (Endocrine disorders) | 18 | 15
Diarrhoea (Gastrointestinal disorders) | 83 | 89
Nausea (Gastrointestinal disorders) | 24 | 40
Stomatitis (Gastrointestinal disorders) | 21 | 31
Vomiting (Gastrointestinal disorders) | 16 | 36
Abdominal pain (Gastrointestinal disorders) | 24 | 27
Constipation (Gastrointestinal disorders) | 20 | 23
Abdominal pain upper (Gastrointestinal disorders) | 19 | 12
Dry mouth (Gastrointestinal disorders) | 17 | 10
Dyspepsia (Gastrointestinal disorders) | 12 | 12
Toothache (Gastrointestinal disorders) | 9 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 8
Haemorrhoids (Gastrointestinal disorders) | 9 | 9
Dysphagia (Gastrointestinal disorders) | 8 | 8
Mouth ulceration (Gastrointestinal disorders) | 5 | 9
Oral pain (Gastrointestinal disorders) | 8 | 6
Fatigue (General disorders) | 43 | 48
Asthenia (General disorders) | 32 | 36
Mucosal inflammation (General disorders) | 23 | 38
Chest pain (General disorders) | 12 | 3
Pyrexia (General disorders) | 4 | 9
Oedema peripheral (General disorders) | 5 | 7
General physical health deterioration (General disorders) | 2 | 8
Urinary tract infection (Infections and infestations) | 9 | 15
Upper respiratory tract infection (Infections and infestations) | 8 | 11
Weight decreased (Investigations) | 38 | 65
Aspartate aminotransferase increased (Investigations) | 35 | 38
Alanine aminotransferase increased (Investigations) | 36 | 36
Blood thyroid stimulating hormone increased (Investigations) | 16 | 21
Gamma-glutamyltransferase increased (Investigations) | 15 | 15
Blood lactate dehydrogenase increased (Investigations) | 11 | 16
Blood alkaline phosphatase increased (Investigations) | 13 | 12
Lipase increased (Investigations) | 13 | 9
Amylase increased (Investigations) | 12 | 8
Blood bilirubin increased (Investigations) | 8 | 9
White blood cell count decreased (Investigations) | 6 | 8
Neutrophil count decreased (Investigations) | 2 | 7
Decreased appetite (Metabolism and nutrition disorders) | 44 | 46
Hypocalcaemia (Metabolism and nutrition disorders) | 31 | 35
Hypomagnesaemia (Metabolism and nutrition disorders) | 16 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 21
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Dysgeusia (Nervous system disorders) | 27 | 23
Headache (Nervous system disorders) | 23 | 18
Dizziness (Nervous system disorders) | 12 | 14
Paraesthesia (Nervous system disorders) | 9 | 6
Insomnia (Psychiatric disorders) | 12 | 10
Proteinuria (Renal and urinary disorders) | 18 | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 67 | 66
Hair colour changes (Skin and subcutaneous tissue disorders) | 22 | 24
Rash (Skin and subcutaneous tissue disorders) | 11 | 22
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 23
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 11
Hypertension (Vascular disorders) | 25 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT01896479/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT01896479/SAP_001.pdf